CLINICAL TRIAL: NCT02371278
Title: Influence of Leucine Co-ingestion With Mixed Meals on Integrative Myofibrillar Protein Synthesis in Older Adults
Brief Title: Leucine Co-ingestion and Myofibrillar Protein Synthesis in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Stuart M. Phillips, Professor Stuart M. Phillips, Ph.D. FACN, FACSM, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LEU-MEALS-2015
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Aging; Sarcopenia
Keywords: Leucine; Protein; Diet; Muscle protein synthesis
MeSH Terms: conditions — Sarcopenia | interventions — Leucine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher daily protein (Other): Diets will provide protein intakes of 1.2 g/kg/d.
  Placebo with meals for 3 days, and leucine with meals for 3 days.
  Interventions: Dietary Supplement: Leucine; Dietary Supplement: Placebo
- Lower daily protein (Other): Diets will provide protein intakes of 0.8 g/kg/d.
  Placebo with meals for 3 days, and leucine with meals for 3 days.
  Interventions: Dietary Supplement: Leucine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Leucine — 5 g leucine with sucrose and maltodextrin
Dietary Supplement: Placebo — 5 g glycine with sucrose and maltodextrin

SUMMARY:
The loss of muscle mass with aging is associated with a dysregulation of muscle protein synthesis (MPS) that is generally characterized by a suppressed MPS response to protein ingestion. This 'anabolic resistance' to protein feeding can be overcome with the ingestion of larger protein servings (~0.4g/kg/meal, equivalent to ~ 30 - 40g/meal); however, older adults would likely find it challenging to consume such quantities of protein on a per meal basis.

The amino acid leucine has a unique role as a key 'activator' of MPS. Some research shows that increasing the leucine content of a suboptimal dose of a protein supplement can enhance the MPS response in older adults. However it is currently unknown whether the co-ingestion of leucine with normal, mixed meals can increase MPS. Furthermore, it has been suggested that leucine supplementation may only benefit older adults consuming suboptimal daily protein intakes. Therefore, the purpose of the current study is to examine the impact of leucine co-ingestion with mixed macronutrient meals on the myofibrillar protein synthetic response in older men consuming daily protein intakes at or below the current recommendations. A further objective is to determine whether the myofibrillar protein synthetic response to a session of resistance exercise is enhanced by leucine supplementation with meals. The investigators hypothesize that, in both the exercised and non-exercised condition, leucine co-ingestion at meals will enhance integrative myofibrillar protein synthesis in older adults consuming lower daily protein intakes, but will not augment MPS in those consuming higher daily protein. The investigators further hypothesize that the influence of leucine supplementation on MPS will be greater in the exercise condition than the non-exercise condition.

DETAILED DESCRIPTION:
At baseline, participants will be asked to wear a pedometer and to complete a physical activity and a weighed food record for 3 days. Resting energy expenditure (indirect calorimetry), body weight and body composition (DEXA) will be assessed in the fasted state. A strength test will be conducted to determine 1 repetition maximum (1-RM) and the maximum load that each participant can lift for 15 - 24 repetitions using a seated leg extension machine. Participants will then be randomized to one of two groups matched for age, activity level and BMI: higher (1.2 g/kg/d) or lower daily protein (0.8 g/kg/d). Participants will then commence a 9 day controlled diet (day -3 to 6) designed to meet energy requirements for weight maintenance and to provide a daily protein intake according to each participant's group allocation (i.e. 0.8 or 1.2 g/kg/d).

All participants will be provided with flavored, supplemental beverages (Infinit Nutrition, Windsor, Ontario) and will be instructed to consume one beverage half way through each meal from day 0 - 5. Individual servings of the supplement will be packaged into a ziplocked pouch by Infinit Nutrition in power form. Participants will be required to add water to the power at home. During day 0 - 2 (unsupplemented period) the beverage will be a placebo (maltodextrin and sucrose), and during day 3 - 5 (leucine supplementation period) the beverage will contain crystalline leucine (5 g) with sucrose for flavour. The beverages will be provided in a single-blind manner, energy-matched and will be similar in odour, color, and taste. Participants will also be blinded to their group allocation.

Aminoacidemia, insulinemia and glycaemia will be determined in response to breakfast, lunch and dinner ingestion during the unsupplemented (day 2) and leucine supplemented (day 5) periods. During each of these blood sampling trials blood samples will be obtained immediately before and 20, 40, 60, 90, 120, 180, 240 min following the ingestion of each meal (total of 25 x 4ml blood samples per participant per trial).

Integrative MPS will be measured in the exercised and non-exercised leg over the unsupplemented (day 0 - 3) period and leucine supplemented (day 3 - 6) period using orally ingested deuterated water (D20) and muscle biopsies obtained from the vastus lateralis on days 0, 3 and 6. Participants will report to the laboratory in the fasted state on day 0 and, following a muscle biopsy from the vastus lateralis and saliva sample, participants will consume a single 100 ml oral bolus of D20 at approximately 0900. Immediately following the D20 bolus participants will perform a bout of unilateral leg extension exercise (3 sets to volitional failure at the maximum load they can lift for 15-24 repetitions (~40-50% 1-RM)). On day 3 participants will perform an identical resistance exercise session with the exception that repetitions will be clamped at the number achieved on day 0. Following both exercise sessions participants will consume their individualized breakfast (with the placebo beverage on day 0 and with the leucine beverage on day 3) in the laboratory before returning home. Bilateral muscle biopsies will be obtained prior to the exercise on day 3 (end of unsupplemented period) and on day 6 (end of leucine supplemented period). Total body water deuterium enrichment can be used as a surrogate for plasma alanine labelling and will be determined from saliva swabs collected by the participant every morning at 0900. Participants will be instructed to not eat or drink anything for 30 min before saliva sampling and samples will be stored in the participant's freezer before their next visit to the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20-35 kg/m2
* Non-smokers

Exclusion Criteria:

* Diabetes mellitus, prediabetes and the metabolic syndrome
* Cardiovascular disease
* Neuromuscular problems or muscle wasting diseases
* Renal disease
* Gastrointestinal disease
* Musculoskeletal conditions such as rheumatoid arthritis or osteoarthritis
* Infectious disease
* Cancer
* Significant body mass loss in the 1 month period prior to the study
* Vegetarianism
* Use of medications known to interfere with muscle metabolism (i.e. beta-blockers, high dose non-steroidal anti-inflammatory drugs, corticosteroids, hormone replacement therapy, antiarrhythmic drugs, warfarin, prescription strength acne medications, oral hypoglycaemic agents and insulin)
* Regular resistance training or daily step counts >9,000 or <3,500

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein fractional synthetic rate | 3 days
  The incorporation of a stable isotope (deuterium) into muscle tissue will allow for the determination of fractional synthetic rate, which is indicative of muscle protein synthesis.

SECONDARY OUTCOMES:
Aminoacidemia in response to daily meals with and without leucine supplementation | 3 days
Glycaemia in response to daily meals with and without leucine supplementation | 3 days
Insulinemia in response to daily meals with and without leucine supplementation | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Murphy CH, Saddler NI, Devries MC, McGlory C, Baker SK, Phillips SM. Leucine supplementation enhances integrative myofibrillar protein synthesis in free-living older men consuming lower- and higher-protein diets: a parallel-group crossover study. Am J Clin Nutr. 2016 Dec;104(6):1594-1606. doi: 10.3945/ajcn.116.136424. Epub 2016 Nov 9. PMID 27935521